CLINICAL TRIAL: NCT07048418
Title: Aesthetic and Functional Self-Assessment Following Rhinoseptoplasty in Patients With Unilateral Cleft Lip and Palate
Acronym: RHINOFENTE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL25_0017
Record Dates: First submitted 2025-06-19; First posted 2025-07-02 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cleft Lip and Cleft Palate
Keywords: rhinoplasty; septoplasty; rhinoseptoplasty; cleft; CLEFT-Q; nasal obstruction
MeSH Terms: conditions — Cleft Lip; Cleft Palate; Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of cleft lip and palate patients who underwent rhinoseptoplasty in childhood or adolescence.
  Interventions: Other: Mailing and completing CLEFT-Q and NOSE questionnaires

INTERVENTIONS:
Other: Mailing and completing CLEFT-Q and NOSE questionnaires — Mailing and completing CLEFT-Q and NOSE questionnaires

SUMMARY:
Secondary rhino-septoplasty in unilateral cleft lip and palate is the treatment of choice for the correction of aesthetic deformities and the functional impact on ventilation nasal. It remains a difficult treatment. It can be proposed at the end of growth or from the age of 10, depending on nasal obstruction and the severity of the deformity.

The CLEFT-Q questionnaire, validated in 2017, has not yet been widely used in studies. The NOSE questionnaire is an older functional questionnaire that is complementary to the CLEFT-Q.

Cleft lip and palate are rare diseases, accounting for around 30% of all facial clefts, which occur at a rate of 1/750 births in Europe. Deformation of the nose and nasal septum is constant, and more or less severe in unilateral forms.

In the absence of rhino-septoplasty performed during primary cleft repair surgery, deformities persist in children and adolescents. There is a significant aesthetic impact in children, which generally increases in adolescents. The problem of nasal obstruction causes functional discomfort that can be disabling. Open rhino-septoplasty is a standard procedure and is proposed as a secondary treatment in this population . It is indicated during growth in cases of nasal obstruction, or as a function of aesthetic demands.

The hypothesis is that secondary rhino-septoplasty gives long-term satisfaction in patients in terms of aesthetics and respiratory function. The originality of this study lies in the use of the recently validated CLEFT-Q questionnaire to assess the aesthetic and functional satisfaction of patients in adulthood after secondary rhino-septoplasty performed in childhood or adolescence. This long-term follow-up will enable us to assess the stability of aesthetic and functional results.

ELIGIBILITY:
Inclusion Criteria:

Unilateral cleft lip and palate Surgery performed at the university hospital as primary surgery (before 12 months of age) without rhino-septoplasty Rhino-septoplasty performed at the university hospital as secondary surgery in childhood or adolescence Aged between 18 and 30 years at the time the CLEFT Q questionnaire was sent out.

Exclusion Criteria:

Incomplete clinical file Primary operation elsewhere than at the Montpellier University Hospital Other operation on the nose prior to rhinoseptoplasty Subject unable to read and/or write Impossibility of following the patient during the study period Opposition to participation after a period of reflection Non affiliation to a social security scheme Persons subject to a legal protection measure (placed under safeguard of justice, persons under guardianship or curatorship), Persons participating in another research study including an exclusion period still in progress Pregnant or breast-feeding women

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Unilateral cleft lip and palate patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Nasal Obstruction and Septoplasty Effectiveness (NOSE) Scale | At inclusion (i.e. 3 to 20 years after surgery, according to inclusion criteria)
  The Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE) consists of 5 items with 5 modalities (from 0 to 4) with higher scores indicating more severe symptoms : nasal congestion, nasal obstruction, difficulty breathing through the nose, sleep disturbance and breathing difficulties during exercise.
CLEFT-Q nose appearance | At inclusion (i.e. 3 to 20 years after surgery, according to inclusion criteria)
  A raw score is first calculated as the sum of the scale items, then rescaled from a conversion table into a score from 0 (worst) to 100 (best).
CLEFT-Q nostrils appearance | At inclusion (i.e. 3 to 20 years after surgery, according to inclusion criteria)
  A raw score is first calculated as the sum of the scale items, then rescaled from a conversion table into a score from 0 (worst) to 100 (best).
CLEFT-Q face appearance | At inclusion (i.e. 3 to 20 years after surgery, according to inclusion criteria)
  A raw score is first calculated as the sum of the scale items, then rescaled from a conversion table into a score from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Asher Mc Dade Score | At least 6 months after surgery
  The aesthetic result is assessed on the basis of photographs (from the medical file) of the face, profile and lower view of the face before/after surgery, using the Asher-McDade method (score from 3 : best appearance to 15 : worst appearance)
Surgical complications according to the Clavien Dindo classification | few days after surgery
  The Clavien-Dindo classification ranges from Grade 1 (minor deviation from normal recovery without pharmacological treatment) to Grade 5 (death). Grade 2 involves complications requiring drugs like antibiotics or blood transfusions. Grade 3 includes complications requiring surgical, endoscopic, or radiological intervention (IIIa without general anesthesia, IIIb with). Grade 4 refers to life-threatening complications needing ICU care (IVa single organ failure, IVb multi-organ). This system standardizes reporting and allows comparison of surgical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided